CLINICAL TRIAL: NCT05326347
Title: A Multicenter, Uncontrolled, Open-label Trial to Investigate the Long-term Tolerability, Safety, and Efficacy of Brexpiprazole Once-weekly (QW) Formulation Administered Once Weekly for 52 Weeks in Patients With Schizophrenia
Brief Title: A Long-term Administration Trial of Brexpiprazole Once-weekly (QW) Formulation in Patients With Schizophrenia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-102-00063
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rollover subjects (Experimental): For rollover subjects, treatment will begin with oral administration of 1 tablet of the brexpiprazole QW formulation at 24 mg. From Week 1 onward, 2 tablets of brexpiprazole QW formulation 24 mg (48 mg/week) will be orally administered for 51 weeks.
  Interventions: Drug: OPC-34712FUM/ Brexpiprazole fumarate
- New subjects (Experimental): In medication switching period, treatment will begin with oral administration of 1 tablet of the brexpiprazole QW formulation 24 mg, and the dose of the other antipsychotics will be gradually reduced, finally switching to monotherapy with 2 tablets of brexpiprazole QW formulation 24 mg (48 mg/week) by Week 4. In treatment period, 2 tablets of brexpiprazole QW formulation 24 mg (48 mg/week) will be orally administered for 52 weeks.
  Interventions: Drug: OPC-34712FUM/ Brexpiprazole fumarate

INTERVENTIONS:
Drug: OPC-34712FUM/ Brexpiprazole fumarate — The treatment will begin with oral administration of 1 tablet of the brexpiprazole QW formulation.

SUMMARY:
Confirm the tolerability and safety of long-term administration of the brexpiprazole QW formulation in patients with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

New Subjects

* Patients who have been fully informed of and understand the objectives, procedures, risks, and expected medicinal benefits of the trial and are able to provide written informed consent prior to initiation of any trial-related procedures
* Patients at least 18 years of age and below the age of 75 at the time of informed consent
* Patients with a diagnosis of schizophrenia based on DSM-5® at the time of informed consent
* Patients who are receiving treatment with antipsychotics (other than clozapine), who are considered to require maintenance therapy using antipsychotics, and for whom monotherapy with the brexpiprazole QW formulation and outpatient management are considered feasible. Hospitalization for washout from any previously used drugs specified as prohibited concomitant drugs or hospitalization for symptom management immediately after the start of IMP administration will be allowed at the discretion of the investigator. Hospitalization for social reasons (eg, homelessness or need for shelter that is unrelated to the patient's psychological condition) is permitted.

Period 1:

- Patients for whom switching to monotherapy with the brexpiprazole QW formulation using an add-on and taper-off method within 4 weeks is considered feasible

Period 2:

* Patients who are able to begin monotherapy with the brexpiprazole QW formulation (at an initial dose of 48 mg/week) Rollover Subjects
* Patients who have been fully informed of and understand the objectives, procedures, risks, and expected medicinal benefits of the trial and are able to provide written informed consent prior to initiation of any trial-related procedures
* Patients who have completed the 6-week double-blind treatment period in Trial 331-102-00062
* Patients for whom monotherapy with the brexpiprazole QW formulation and outpatient management are considered feasible. Hospitalization for symptom management immediately after the start of IMP administration will be allowed at the discretion of the investigator. Hospitalization for social reasons (eg, homelessness or need for shelter that is unrelated to the patient's psychological condition) is permitted.

Exclusion Criteria:

New Subjects

* Patients who are considered resistant/refractory to antipsychotic treatment Patients who are
* Patients who are considered resistant/refractory to antipsychotic treatment Patients who are "unresponsive to medication with 2 or more antipsychotics at effective doses for a sufficiently long duration (6 weeks)" will be deemed resistant/refractory to antipsychotic treatment.
* Patients experiencing acute depressive symptoms within 30 days prior to informed consent that, in the judgment of the investigator, require treatment with an antidepressant
* Patients who fall under any of the following criteria regarding suicidal ideation and suicidal behavior

  1. Patients who answered "yes" to Question 4 "Active Suicidal Ideation with Some Intent to Act, without Specific Plan" or Question 5 "Active Suicidal Ideation with Specific Plan and Intent" regarding Columbia-Suicide Severity Rating Scale (C-SSRS) suicidal ideation at screening (for the past 6 months) or at baseline (since the last assessment)
  2. Patients who exhibited suicidal behavior on C-SSRS at screening (for the past 2 years) or at baseline (since the last assessment)
  3. Patients who present a serious risk of suicide based on the judgment of the investigator
* Patients presenting tardive dyskinesia at the time of informed consent, as determined by a score of 3 (moderate) or 4 (severe) for Item 8 (severity of abnormal movements) of the Abnormal Involuntary Movement Scale (AIMS) at screening or at baseline
* Patients with a score of 5 (severe akathisia) in the Barnes Akathisia Rating Scale (BARS) global clinical assessment of akathisia at screening or at baseline
* Patients with a diagnosis of a concurrent mental disorder besides schizophrenia (schizoaffective disorder, major depressive disorder, bipolar I disorder, bipolar II disorder, general anxiety disorder, obsessive-compulsive disorder, post-traumatic stress disorder, dementia or mild neurocognitive disorder, personality disorder, etc) based on DSM-5®. However, this exclusion does not apply to the following:

  • Caffeine- or tobacco-related disorder
* Patients who have met the DSM-5® diagnostic criteria for substance-related or addictive disorder, including alcohol and benzodiazepines but excluding caffeine and tobacco, within 180 days before commencement of IMP administration
* Patients who have a clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorder. Medical conditions that are minor or well-controlled may be c+E97onsidered acceptable if the condition does not interfere with safety and efficacy assessments.
* Patients with known hypersensitivity or intolerance to brexpiprazole or patients with confirmed resistance to brexpiprazole therapy
* Patients judged by the investigator to be unsuitable for participation in the trial Rollover Subjects
* Patients who have a clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorder. Medical conditions that are minor or well-controlled may be considered acceptable if the condition does not interfere with safety and efficacy assessments.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The frequency of Adverse Events | From baseline to week 52

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Tsunoda, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Hayakawa Clinic, Kure-shi, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.